CLINICAL TRIAL: NCT02988206
Title: Personalized Objects Can Improve the Diagnosis of EMCS From MCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Yuxiao Sun, Undergraduate student, Hangzhou Normal University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2016R423055
Record Dates: First submitted 2016-12-05; First posted 2016-12-09 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Patients in Minimally Conscious State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalized Objects (Other): The item "Functional Object Use" was assessed by using personalized objects (e.g., cigarette, paper) and non-personalized objects, which presented in a random order..
  Interventions: Behavioral: Personalized Objects; Behavioral: non-personalized Objects
- non-personalized objects (Other): The item "Functional Object Use" was assessed by using non-personalized objects
  Interventions: Behavioral: non-personalized Objects

INTERVENTIONS:
Behavioral: Personalized Objects — personalized objects are based on the observation or the reports from family
  Arms: Personalized Objects
Behavioral: non-personalized Objects — non-personalized objects are based on the suggestion in CRS-R,which are comb and cup

SUMMARY:
In this study，researchers will use personalized objects to assess patients' level of consciousness in chronic patients in minimally conscious state (MCS).

DETAILED DESCRIPTION:
The Coma Recovery Scale-Revised (CRS-R) is an important tool for the assessment of behaviors in DOC.Clinical practice has shown that self-referential stimuli, such as the patient's own name and face, are more effective to elicit the patient's response than that of non-self-referential stimuli.

The item "Functional Object Use" was assessed by using personalized objects (e.g., cigarette, paper) and non-personalized objects, which presented in a random order.The rest assessments were performed following the standard protocol of CRS-R. The differences between functional use of the two types of objects was analyzed by Chi-square test.

Researchers expected to see some of the patients in MCS are re-diagnosed as EMCS with the using of personalized objects.

ELIGIBILITY:
Inclusion Criteria:

* patients in minimally conscious state;
* patients with stable condition;
* each patient has athletic ability to some extent.

Exclusion Criteria:

* premorbid neurology antecedent;
* patients in coma or vegetative state;
* patients < 1 months after the acute brain injury.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The frequency of behavioral response elicited by the stimuli suggested by CRS-R scale and the personalized stimuli they prefer | one week

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun Y, Wang J, Heine L, Huang W, Wang J, Hu N, Hu X, Fang X, Huang S, Laureys S, Di H. Personalized objects can optimize the diagnosis of EMCS in the assessment of functional object use in the CRS-R: a double blind, randomized clinical trial. BMC Neurol. 2018 Apr 12;18(1):38. doi: 10.1186/s12883-018-1040-5. PMID 29649978